CLINICAL TRIAL: NCT05188950
Title: Effectiveness of a Cognitive Behavioral Therapy Based Mobile Application in College Students With Depression Symptoms
Brief Title: Effectiveness of a CBT Based Mobile Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Yuanpei University of Medical Technology (Other); Fooyin University (Other); Tajen University (Unknown); Taiwan Nurses Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 202108098RINB
Record Dates: First submitted 2021-12-08; First posted 2022-01-12 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2021-10

CONDITIONS: Depressive Symptoms
Keywords: mobile application; cognitive behavioral therapy; depression symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): The intervention involved the participants' use of the mobile application.
  Interventions: Device: depression screening test App
- control group (No Intervention): As usual.

INTERVENTIONS:
Device: depression screening test App — The participants' use of the depression screening test App of 6 modules for 12 weeks, at least once a week, 20 minutes per once.
  Arms: treatment group

SUMMARY:
This research aims to explore the effect of a mobile application designed on the basis of cognitive behavioral therapy on college students suffering from depression in terms of their symptoms, suicidal thoughts, and other relevant variables.

DETAILED DESCRIPTION:
Background: College students encounter the transition from adolescence to adulthood, thereby possibly facing various factors causing depression. However, instead of consulting a professional, most college students seek help online or through contacts, or internalize their emotions. The current situation could be due to the low efficiency of depression prevention and the limited consultation provided at campus. While many studies have examined adopting mobile applications in dealing with depression, they have not shown consistent results. The cross-sectional research has been the most common; few randomized controlled trials have been conducted. Hence, much empirical evidence is needed to identify the effect of a mobile application.

Aim: This research aims to explore the effect of a mobile application designed on the basis of cognitive behavioral therapy on college students suffering from depression in terms of their symptoms, suicidal ideation, and other relevant variables.

Methodology: This is a randomized controlled trials study. The participants, aged 20 and above, were recruited from three universities of science and technology of similar nature. All of them suffer from depression symptoms and have used Wi-Fi smartphones. They were randomly assigned to the control group and the treatment group. The treatment group received an intervention involving the participants' use of the mobile application for 12 weeks, at least once a week, 20 minutes per session. The generalized estimating equation was adopted to analyze the results regarding the depression symptoms, suicidal ideation, help-seeking attitudes, emotional self-awareness, and mobile health (mHealth) literacy.

Expected outcomes: The results obtained by tracking the symptoms of depression from the empirical research design conducted on campus will provide a reference to understanding to what extent mobile applications could be an appropriate intervention for college students.

Clinical application: The research findings could provide insights for policymaking in respect of helping a person with depression on campus to better meet college students' needs.

ELIGIBILITY:
Inclusion Criteria:

* suffer from depression symptoms.
* aged 20 and above.
* being able to communicate in Chinese or Taiwanese.
* used Wi-Fi smartphones.
* Agree and obtain written consent.
* In the school term during research.

Exclusion Criteria:

* Have a full-time job.
* Who has been diagnosed with bipolar disorder, Asperger syndrome, and schizophrenia.
* Who have the health conditions associated with visual impairments, auditory impairments, and mobility impairments, that are limited to the use of accessibility mobile applications.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Change from baseline (1st week) in depressive symptoms on the Tung's Depression Inventory for College Students (TDICS) at Week 4, 8,12. | Baseline(1st week) and 4th week, 8th week,12th week.
  The Tung's Depression Inventory for College Students (TDICS) is validated. It comprised of 32 items in 4-point Likert-type format and can be completed between 5 to 10 minutes. The scores range from 0 (no depressive) to 96 (high depressive symptoms).
Change from Baseline(1st week) in suicide ideation on Concise Mental Health Checklist (CMHC) at Week 4, 8,12. | Baseline(1st week) and 4th week, 8th week,12th week.
  The Concise Mental Health Checklist (CMHC) is validated. The scores range from 0 (no suicide ideation) to 9 (high suicide ideation).

SECONDARY OUTCOMES:
Change from Baseline(1st week) in emotional self-awareness on Emotional Self-Awareness Scale - Revised (ESAS-R) at Week 4, 8,12. | Baseline(1st week) and 4th week, 8th week,12th week.
  Emotional Self-Awareness Scale - Revised (ESAS-R) is validated. The scores range from 0 (no emotional self-awareness) to 84 (high emotional self-awareness).
Change from Baseline(1st week) in help-seeking attitudes on Attitudes Toward Seeking Professional Psychological Help Shortened Form (ATSPPH-SF) at Week 4, 8,12. | Baseline(1st week) and 4th week, 8th week,12th week.
  The Attitudes Toward Seeking Professional Psychological Help Shortened Form (ATSPPH-SF) is validated. The scores range from 0 (low help-seeking attitudes) to 30 (positive help-seeking attitudes).
Change from Baseline(1st week) in mHealth literacy on mHealth literacy of app Scale at Week 4, 8,12. | Baseline(1st week) and 4th week, 8th week,12th week.
  The mHealth literacy of app Scale is development by YHL researcher. The purpose of the scale was to develop a screening tool for mHealth literacy of app. Only the treatment group needs to fill this instrument. It is comprised of 8 items in 5-point Likert-type format. The scores range from 8 (low mHealth literacy of app) to 40 (high mHealth literacy of app).

CONTACTS AND LOCATIONS:
Overall Officials: Meei-Fang Lou, Ph.D., Principal Investigator — School of Nursing, College of Medicine, National Taiwan University
Locations (1):
- School of Nursing, College of Medicine, National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data.

REFERENCES:
- [Derived] Lin YH, Wu CY, Gau BS, Lin CH, Ho HY, Lou MF. Effectiveness Study of a Cultural Adaptation of Cognitive-Behavioural Therapy-Based Application for Depressive Symptoms in College Students: A Randomised Controlled Trial. J Psychiatr Ment Health Nurs. 2025 Jun;32(3):712-722. doi: 10.1111/jpm.13146. Epub 2024 Dec 18. PMID 39692262